CLINICAL TRIAL: NCT05522777
Title: Survival of the Probiotic Lacticaseibacillus Paracasei Strain Shirota (LcS) in the Gastrointestinal Tract of Generally Healthy Adults
Brief Title: Survival of the Probiotic Lacticaseibacillus Paracasei Strain Shirota (LcS) in the GI Tract of Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult U.S.A. Inc. (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry); Illinois Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BIO-2208
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: probiotics; Lacticaseibacillus paracasei strain Shirota; Colony Forming Unit; survival in GI tract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product consumption group (Experimental): Drink one bottle of Yakult a day
  Interventions: Other: Drink one bottle of Yakult a day

INTERVENTIONS:
Other: Drink one bottle of Yakult a day — Yakult is a branded probiotic drink with 8x10^9 CFU Lacticaseibacillus paracasei strain Shirota

SUMMARY:
The objective of this study is to investigate the survival of Lacticaseibacillus paracasei strain Shirota (LcS) in the human gastrointestinal (GI) tract after consumption of probiotics fermented milk product containing 8x10^9 LcS. This study is a single-arm, open-label study with a 14-d run-in (baseline), 14-d consumption period, and 14-d follow-up. Participants will maintain habitual dietary and lifestyle practices with the exception of avoiding fermented foods and beverages throughout the 42-d trial. The number of live LcS in fecal samples will be assessed after 14 d consumption of a fermented milk product.

DETAILED DESCRIPTION:
The study is a single-arm, open-label study with one screening visit (Visit 1; Day 0), one baseline visit (Visit 2; Day 14), two intervention visits (Visits 3 and 4; Days 21 and 28), and one post-intervention follow-up visit (Visit 5; Day 42).

After signing the informed consent, participants will be screened for eligibility. All women will be required to take an in-clinic urine pregnancy test. After review of inclusion/ exclusion criteria, eligible participants will then be enrolled in the study and start a 14-d run-in period. Eligible participant will be instructed to continue with their habitual diets and lifestyle patterns, with exception of excluding fermented dairy and non-dairy products. A Stool Collection Demonstration will be conducted and participants will be provided a stool collection kit, along with ice packs. Participants will be instructed to collect a stool sample sometime after 7 pm the day before and prior to their next visit (Visit 2; Day 14). Participants will also be instructed on the electronic Daily Diary, which asks compliance with study instructions to avoid fermented products as well as questions on concomitant medication intake. Visit 2 (Day 14) is the end of the run-in and start of the ingestion period. At Visit 2, participants will arrive in the morning, undergo clinic procedures. Stool samples will be collected (Day 14 samples), and the eDiaries reviewed as appropriate. Additionally, participants will be queried about following the study instructions provided at Visit 1. The first serving of study product will be consumed during the clinic visit after participants have consumed breakfast (at home) and obtained and dropped off their stool samples. Participants will then be dispensed two 5-packs of study product for at-home daily consumption until the next visit (Visit 3; Day 21) and instructed to consume one bottle of the study product within the 30 minutes following breakfast, and to keep all dispensed product refrigerated prior to consumption. A new stool collection kit with fecal sample storage materials will be provided and participants instructed to collect a stool sample sometime after 7 pm the day before and prior to their next visit (Visit 3; Day 21). Participants will be reminded to maintain their habitual dietary and lifestyle patterns and refrain from consumption of any other fermented dairy and non-dairy products, consume their study product daily, and complete their eDiaries every day. The eDiary will contain the same questions as during the run-in plus queries on daily product consumption, which will then be used for compliance assessment. Adverse events (AE) will be assessed by open-ended question at the beginning and end of Visit 2 (Day 14) and at the beginning of Visits 3, 4, and 5 (Days 21, 28, and 42, respectively). Participants will be counseled to contact the clinic with concerns or discomforts. If participants miss consuming study product in the morning, they should be counseled to consume the product as soon as possible during that day; however, participants should not consume more than one serving of product per day. Therefore, if they miss consuming the product during the entire day, they should document the lack of study product consumption and continue consuming one serving per day. Following the first seven days of the ingestion period, participants will return for an interim visit (Visit 3; Day 21) to drop off their stool sample (Day 21 sample) and to obtain a new stool collection kit. Participants will be instructed to collect another stool sample (Visit 4; Day 28). The eDiary will be reviewed, including product consumption compliance, and participants will be queried about following the study instructions. AEs will be assessed. Participants will return unused study product and be dispensed new study product to continue at-home daily consumption, with reminder to consume one serving per day until the next visit. Participants will also be reminded to continue to maintain habitual dietary and lifestyle patterns while avoiding fermented dairy and non-dairy products, as well as to complete their eDiaries every day. At the end of the ingestion period, participants will return for Visit 4 (Day 28) to drop off their stool sample (Day 28 sample) and return unused study product. Clinic procedures will be performed, AEs assessed, and electronic Daily Diaries and compliance will be reviewed. At this point, participants will be instructed that will no longer need to consume study product and will enter the follow-up period. Participants will be dispensed a new stool collection kit and instructed to collect a final stool sample (Visit 5; Day 42). Participants will also be reminded to continue to maintain habitual dietary and lifestyle patterns while avoiding fermented dairy and non-dairy products as well as to complete their eDiaries every day. Participants will return for their final visit (Visit 5; Day 42) after collection of their follow-up stool sample (Day 42 sample). Participants will drop off their final stool sample. Clinic visit procedures will be conducted, AEs assessed, and participants will be queried about following study instructions. eDiaries will be reviewed as appropriate. Participants will then be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18-40 years old, inclusive at Visit 1.
2. BMI between ≥18.5 to ≤29.9 kg/m2.
3. Regular bowel habits, by self-report, including consistently having a bowel movement every day, preferably in the morning.
4. Regular breakfast consumer by self-report.
5. Willing to consume the study product per the protocol instructions throughout the study intervention period (14 d).
6. Willing to maintain habitual dietary, lifestyle, and physical activity (with exceptions per study instructions) throughout the trial and to refrain from exclusionary medications, supplements, and products throughout the study.
7. Willing to limit alcohol consumption to ≤3 standard drinks/d and ≤7 standard drinks/wk throughout the trial.
8. Non-user of tobacco products or former user of any tobacco product (not used within 6 months) and has no plan to change nicotine habits during the study period. Tobacco products include tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 6 months of Visit 1 (Day 0) and during the study period.
9. Non-user or former user of any marijuana or hemp products (not used within 6 months) of Visit 1 (Day 0) and during the study period and has no plans to use marijuana or hemp products during the study period. No washout is required for topical marijuana or hemp products, but subjects are required to abstain from these products during the study period.
10. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Any known food allergies, intolerances or sensitivities to dairy or to any of the study product ingredients.
2. Presence of a clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies). IBS will be determined as recurrent abdominal pain or discomfort at least 3 d/mo in the last 3 mo associated with: (a) improvement with defecation, (b) onset associated with change in frequency of stool, and (c) onset associated with a change in form (appearance of stool).
3. Self-reported history (within 6 wks) or presence of functional constipation or diarrhea as defined by the Rome IV criteria and at the discretion of the Clinical Investigator.

   * Diarrhea is defined as loose or watery stools, without predominant abdominal pain or bothersome bloating, occurring in more than 25% of stools.
   * Constipation is defined as two or more of the following: (a) straining during more than ¼ (25%) of defecations; (b) lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations; (c) sensation of incomplete evacuation more than ¼ (25%) of defecations; (d) sensation of anorectal obstruction/blockage more than ¼ (25%) of defecations; (e) manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor); (f) fewer than 3 single bowel movements/ per week; (g) loose stools are rarely present without the use of laxatives.
4. Self-reported history (within 6 wks) or presence of abdominal pain, defined as continuous or nearly continuous pain in the abdominal area in which (a) no or only occasional relationship with physiological events (e.g., eating, defecation, menses), (b) some loss of daily functioning (pain limits activity at least some of the time), (c) the pain is not feigned, (d) the pain is not related to another GI disorder (e.g., epigastric pain syndrome, irritable bowel syndrome, anorectal pain).
5. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), hepatic, renal (except history of kidney stones in participants who are symptom free for 6 months), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary condition(s). Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day 0). One re-test may be allowed on a separate day prior, with repeating of Visit 1, for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Day 0), in the judgment of the Clinical Investigator. If taken, the repeat blood pressure measurement will be used to determine eligibility. Stable use of hypertension medication is allowed [defined as no change in medication regimen within 90 d of Visit 1 (Day 0)].
7. Weight loss or gain > 4.5 kg within 90 d of Visit 1 (Day 0), or currently or planning to be on a weight loss regimen or muscle-building/strengthening program during the study.
8. Signs or symptoms of an active infection of clinical relevance within 5 d of Visit 1 (Day 0). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 d prior to Visit 1 (Day 0).
9. Major trauma or any other surgical event within 90 d of Visit 1 (Day 0).
10. History or presence of cancer in the prior 2 y, except for non-melanoma skin cancer.
11. Use of proton pump inhibitors, H2 receptor antagonists, anticoagulants (with the exception of 81 mg aspirin), corticosteroids, antibiotics, antifungals, antiparasitics, antidiarrheals, laxatives, or regular (> 3 d/wk) use of NSAIDs within 30 d of Visit 1 (Day 0).
12. Exposure to any non-registered drug product within 30 days prior to Visit 1 (Day 0).
13. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception during the study period. The method of contraception must be recorded.
14. Recent history (within 12 mo of screening; Visit 1; Day 0) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks/wk (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
15. Recent (within 2 mo) participation in any other clinical study prior to Visit 1 (Day 0).
16. Has a condition the Clinical Investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

    -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Yakult U.S.A. Inc, Fountain Valley, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew at the baseline visit due to schedule conflict.
Period: Overall Study
Arm/Group | Test Product Consumption Group
Started | 26 (One participant withdrew before starting ingestion period, so one additional participant was recruited and enrolled.)
Completed | 24
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test Product Consumption Group
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.0 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Live LcS Numbers From Baseline (Day 14) to the End of the Ingestion Period (Day 28).
Description: The change in Live LcS numbers (CFU/g Feces) from baseline (Visit 2; Day 14) to the end of the ingestion period (Visit 4; Day 28) was measured by colony PCR method.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: Log 10 CFU/g Feces
Arm/Group | Test Product Consumption Group
Number analyzed (Participants) | 24
Log 10 CFU/g Feces
  Number of LcS at Day 14 | 2.14 [1.89 to 2.44]
  Number of LcS at Day 28 | 5.27 [4.50 to 6.04]

2. Secondary Outcome: Change in LcS Number From Baseline (Day 14) to the Mid of Ingestion Period (Day 21).
Description: The change in Live LcS numbers (CFU/g Feces) from baseline (Visit 2; Day 14) to the mid of ingestion period (Visit 3 ; Day 21) was measured by colony PCR method.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: Log10 CFU/g feces
Arm/Group | Test Product Consumption Group
Number analyzed (Participants) | 24
Log10 CFU/g feces
  Number of LcS at Day 14 | 2.17 [1.89 to 2.44]
  Number of LcS at Day 21 | 6.37 [5.88 to 6.86]

3. Secondary Outcome: Change in LcS Numbers From the End of the Ingestion Period (Day 28) and to the End of Follow-up (Day 42).
Description: The change in LcS numbers from the end of the ingestion period (Visit 4; Day 28) to the end of follow-up period (Visit 5; Day 42) was measured by colony PCR method..
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: Log 10 CFU/g feces
Arm/Group | Test Product Consumption Group
Number analyzed (Participants) | 24
Log 10 CFU/g feces
  Number of LcS at Day 28 | 5.27 [4.50 to 6.04]
  Number of LcS at Day 42 | 2.14 [1.93 to 2.35]

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Test Product Consumption Group
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to disclose the data relating to or the results of the Study to any third party, except as otherwise agreed to in writing by Sponsor for a period of three (3) years from the date the last clinic visit is completed by a Research Subject.

DOCUMENTS (2):
  • Study Protocol (2022-07-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT05522777/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT05522777/SAP_001.pdf